CLINICAL TRIAL: NCT01121380
Title: A First-in-Human, Randomized, Double-Blind, Placebo Controlled, Single-Center Combined Single-Ascending Dose and Multiple-Ascending Dose, Parallel Groups, Study to Assess Safety, Tolerability and Pharmacokinetics of BL-1021 in Healthy Volunteers
Brief Title: A Study Intended to Evaluate Safety, Tolerability and Pharmacokinetics (PK) Parameters of BL-1021
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor strategy change
Sponsor: BioLineRx, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: BL-1021.01
Record Dates: First submitted 2010-05-10; First posted 2010-05-12 (Estimated); Last update posted 2014-03-13 (Estimated); Status verified 2014-03

CONDITIONS: Healthy; Volunteers
Keywords: Healthy; Volunteers

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (8):
- Cohort A - 10 mg (Experimental)
  Interventions: Drug: BL-1021; Drug: 1021
- Cohort B - 20 mg (Experimental)
  Interventions: Drug: BL-1021; Drug: 1021
- Cohort C - 40 mg (Experimental)
  Interventions: Drug: BL-1021; Drug: 1021
- Cohort D - 80 mg (Experimental)
  Interventions: Drug: BL-1021; Drug: 1021
- Cohort E - X mg (Experimental): Part 2, multiple dose. X shall be determined using the results of part 1.
  Interventions: Drug: BL-1021; Drug: 1021
- Cohort F - 2X mg (Experimental): Part 2, multiple dose. X shall be determined using the results of part 1.
  Interventions: Drug: BL-1021; Drug: 1021
- Cohort G - 4X mg (Experimental): Part 2, multiple dose. X shall be determined using the results of part 1.
  Interventions: Drug: BL-1021; Drug: 1021
- Placebo (Placebo Comparator): In each cohort there is a placebo arm
  Interventions: Drug: 1021

INTERVENTIONS:
Drug: BL-1021 — BL-1021 is an orally available NCE which contains an elongated aliphatic side-chain.
  Dosage:
  Part 1 - Single Dose: 1 dose on Day 1, dosage will be 10, 20, 40 & 80 mg according the cohort Part 2 - Multiple Dosing: up to 7 once-daily administrations. Dosage will be determined according the first part results.
  Arms: Cohort A - 10 mg; Cohort B - 20 mg; Cohort C - 40 mg; Cohort D - 80 mg; Cohort E - X mg; Cohort F - 2X mg; Cohort G - 4X mg
Drug: 1021 — 1021

SUMMARY:
The purpose of this study is to test the safety, tolerability and pharmacokinetics of BL-1021 in healthy volunteers. Subsequent clinical studies will be designed to test the safety and efficacy of BL-1021 in patients with neuropathic pain based on data obtained from the proposal trial described below.

DETAILED DESCRIPTION:
A total of 32 subjects in the single-ascending phase and 24 subjects in the multiple ascending phase, who have provided a written informed consent and comply with inclusion/exclusion criteria will participate in the study in 4 different cohorts in the first phase (cohorts A, B, C and D) and 3 different cohorts in the second phase (cohorts E, F and G), each consisting of 8 subjects.

First part dosing:

Cohort A - 10 mg Cohort B - 20 mg Cohort C - 30 mg Cohort D - 40 mg

Second part dosing:

Cohort E - X mg (X shall be determined using the results of the 1st part) Cohort F - 2X mg Cohort G - 4X mg

ELIGIBILITY:
The inclusion criteria for both parts 1 and 2 of the study are:

* Ability to provide written informed consent
* Healthy male between 18 and 45 years of age, inclusive
* BMI of 18-30, inclusive
* Negative urinary drugs of abuse screen within 21 days of start of study
* No significant abnormal blood hematology and biochemistry tests according to the opinion of the principal investigator
* Only subjects with a known (pre-study) CYP2D6 genotype will be enrolled.
* No concomitant medications (prescription, OTC, vitamins, dietary supplements) within 7 days prior to administration of study medication
* Non-smoking (by declaration) for a period of at least 6 months prior to enrolment
* Ability to adhere to the visit schedule and protocol requirements and be available to complete the study
* No significant abnormalities in physical examination

Exclusion criteria for both parts 1 and 2 of the study are:

* Evidence or history of significant concomitant disease (including mental, CNS-related, renal, hepatic, cardiovascular, pulmonary disease, or other)
* Prior or current history of cancer, except for cured basal cell carcinoma of the skin
* History of significant abnormalities in ECG, including QT prolongation
* History of significant neurological, renal, cardiovascular, respiratory (asthma), endocrinological, gastrointestinal, hematopoietic disease, neoplasm (especially melanoma), or any other clinically significant medical disorder, which in the Investigator's judgment contraindicate administration of the study medications
* Use of another investigational medication/treatment in the past 30 days
* History of drug or alcohol abuse
* Significant abnormalities in screening physical examination
* Significant abnormalities in clinical laboratory parameters (hematology, biochemistry, serology, urinalysis)
* History of gastrointestinal disorder likely to influence drug absorption
* Consumption of Serotonin-Norepinephrine Reuptake Inhibitors (SNRI's), selective serotonin reuptake inhibitors (SSRI's), tricyclic/tetracyclic antidepressants within 90 days prior to Day 0
* Consumption of drugs that may potentially inhibit or induce liver cytochrome P450 activity within 3 weeks prior to Day 0
* Subjects who are either extensive-extensive metabolizers (i.e. carriers of multiple CYP2D6 gene copies) or poor metabolizers of CYP 2D6 will be excluded.
* Any acute medical situation (e.g. acute infection) within 48 hours of Day 0, which is considered of significance by the Principal Investigator
* Unusual diet
* Sero-positive HIV, HBSAg or HCV
* Donation of 450ml or more blood within the previous 12 weeks
* Probability of undertaking intense physical activity throughout the study duration (Single Dose: Day 0 - Day 8, Multiple Dose: Day 0 - Day 14)
* Any condition, which in the opinion of the Principal Investigator would place the subject at risk or influence the conduct of the study or interpretation of results
* Inability to communicate well with the Investigator (i.e., language problem, poor mental development or impaired cerebral function)
* Subjects who, in the judgment of the investigators, are likely to be non-compliant or uncooperative or unwilling to sign a consent form

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2011-06; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | Part 1 and 2

SECONDARY OUTCOMES:
Mean change from baseline in vital signs | Part 1 and 2
Mean change from baseline in laboratory parameters | Part 1 and 2
Cmax, Tmax, AUCT, AUCI, kel, T½ | Part 1 and 2
Dose linearity of PK parameters | part 1 and 2

CONTACTS AND LOCATIONS:
Overall Officials: Yotam Nisemblat, Study Director — BioLineRx, Ltd.; Yoseph Caraco, Prof, MD, Principal Investigator — Hadassah Clinical Research Center (HCRC)
Locations (1):
- Hadassah Clinical Research Center (HCRC), Jerusalem, Israel